CLINICAL TRIAL: NCT02018653
Title: A Double-Blinded Placebo-Controlled Pilot Trial of Calcium Alumina-Silicate (CASAD) in the Treatment of Severe Diarrhea (Grade 3 or 4) in Cancer Patients Presenting for Emergency Care
Brief Title: CASAD for Severe Diarrhea in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Salient Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0452; NCI-2014-01027 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Diarrhea
Keywords: Cancer; Diarrhea; Calcium Alumina-Silicate; CASAD; Calcium Aluminosilicate anti-diarrheal; Placebo; Sugar pill; Questionnaire; Survey
MeSH Terms: conditions — Neoplasms; Diarrhea | interventions — Calcium Aluminosilicate; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium Alumina-Silicate (CASAD) (Experimental): CASAD 1 gram orally every 6 hours for up to 6 days. Questionnaire completion at baseline about diarrhea and other symptoms.
  Interventions: Drug: Calcium Alumina-Silicate (CASAD); Behavioral: Questionnaire
- Placebo (Placebo Comparator): Placebo orally every 6 hours for up to 6 days. Questionnaire completion at baseline about diarrhea and other symptoms.
  Interventions: Other: Placebo; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Calcium Alumina-Silicate (CASAD) — 1 gram by mouth every 6 hours for up to 6 days.
  Other Names: CASAD; Calcium Aluminosilicate anti-diarrheal
  Arms: Calcium Alumina-Silicate (CASAD)
Other: Placebo — 1 by mouth every 6 hours for up to 6 days.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Questionnaire — Questionnaire completion at baseline about diarrhea and other symptoms.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if calcium alumina-silicate (CASAD) can help to stop your diarrhea. Researchers also want to know if this drug can help decrease the duration of your diarrhea.

In this study, CASAD will be compared to a placebo. A placebo is not a drug. It looks like the study drug but it is not designed to treat any disease or illness. It is designed in this study to be compared with the study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to receive either CASAD orally or a placebo. You will have an equal chance of being assigned to either group.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Treatment:

You take either CASAD or placebo by mouth every 6 hours with about 1 cup (8 oz.) of water. You will also be given other supportive care and treatment for diarrhea (such as imodium and lomotil).

You will be asked to keep a journal, which includes a record of the time you take the study drug each day and a history of your bowel movements every day you take CASAD or placebo.

Study Visits:

Before the dose:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be recorded.
* You will be asked when your diarrhea started.
* You will be asked about any drugs you have taken for the cancer and diarrhea.
* A stool sample will be collected to test for toxins.
* Blood (about 1 teaspoon) will be drawn to measure cytokines (proteins that may affect the immune system and inflammation) .
* You will be asked about your diarrhea and other symptoms. It should take about 5 minutes to answer these questions.

At the same visit after the dose:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about your diarrhea.
* You will be asked if you have any side effects.

On Day 1 (the day after your visit to the Emergency Center):

-Blood (about 1 teaspoon) will be drawn to check your electrolytes and to measure cytokines and inflammation (optional).

On Days 2-6 (this will be by phone or the staff will visit you if you are in the hospital):

* You will be asked about your diarrhea.
* You will be asked if you have any side effects.

Length of Treatment:

You will take the study drug or placebo for up to 6 days or when the diarrhea stops, whichever happens first. You will no longer be able to take the study drug or placebo if the diarrhea gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Follow-Up:

After you are off study, the study nurse will call you and ask if you have had any other side effects since finishing the study treatment. The phone call should only last about 5 minutes. If you are still an inpatient at the hospital, the study nurse may visit you and ask you these questions in person.

At your next scheduled appointment at MD Anderson, the nurse will meet with you to get your final journal and any unused study drug. If you do not return to MD Anderson, you will receive a self-addressed stamped envelope for you to return this information.

This is an investigational study. CASAD is FDA approved as a food additive, but it has not been approved to treat a disease. Its use to treat diarrhea is investigational.

Up to 24 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients presenting to the EC or an acute care clinic for NCI grade >/= 2 diarrhea
2. Able to understand the description of the study and give informed consent
3. Patients must be willing to and capable of providing frequent assessments for the duration of the study
4. English-speaking

Exclusion Criteria:

1. Patients will not be approached while they have : a) evidence of fever or severe abdominal pain, melena, overt blood in stool; b) any clinical suspicion or evidence of peritonitis or bowel perforation; c) s/p allogenic stem cell transplant
2. Patients will not be approached if the EC physician thinks that the diarrhea is due to Crohn's disease, ulcerative colitis, Celiac disease, graft-versus-host disease, short-gut syndrome, neuroendocrine paraneoplastic syndromes (e.g., MEN, VIPomas, etc.), or malabsorption syndromes
3. Patients who are status post stem cell transplantation (both autologous or allogenic)
4. Patients who are status post immunotherapy (including those who are receiving or have received ipilimumab)
5. Patients participating in other clinical trials for diarrhea
6. Patients with a known allergy to any components of the CASAD formulation
7. Patients whose current medication schedule would not permit an approximate 2 hour window between administration of CASAD and other scheduled medications
8. Patients who cannot comply with medications
9. Patients taking any clay products
10. Patients with radiological evidence of megacolon, intraperitoneal free air, pneumatosis intestinalis, or fecal impaction
11. History of significant neurological or psychiatric disorders that would impede giving consent, treatment, or follow up
12. Patients who are pregnant
13. Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sai-Ching J. Yeung, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 16, 2013 to August 1, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Clinical trial closed due to slow accrual.
Groups:
- Calcium Alumina-Silicate (CASAD): CASAD 1 gram orally every 6 hours for up to 6 days.
- Placebo: Placebo orally every 6 hours for up to 6 days.
Period: Overall Study
Arm/Group | Calcium Alumina-Silicate (CASAD) | Placebo
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Alumina-Silicate (CASAD) | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Diarrhea (TTRD)
Description: The primary endpoint is time to resolution of diarrhea (TTRD) defined as the time of the bowel movement that is not followed by another bowel movement within 8 hours. Participants will be evaluated for the primary endpoint for up to 6 days.
Time Frame: 6 days
Population: Too few subjects enrolled to make any conclusions.
Measure: Number; unit: hours
Arm/Group | Calcium Alumina-Silicate (CASAD) | Placebo
Number analyzed (Participants) | 1 | 1
hours | 48 | 96

ADVERSE EVENTS:
Time Frame: Adverse event monitoring and reporting will begin after participants receive the study drug or placebo and will continue to be recorded through discharge from study, anticipated to be day 6.
Arm/Group | Calcium Alumina-Silicate (CASAD) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes